CLINICAL TRIAL: NCT07267559
Title: An Investigation of the Effects of Dual Orexin Antagonism on Emotional Processing and Learning in Healthy Individuals
Brief Title: Dual Orexin Antagonism and Emotion and Affective Processing Study
Acronym: DOREA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DOREA
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Learning; Cognitive Functioning; Emotional Processing
Keywords: Drug; Orexin; Hypocretin; Healthy volunteers; Learning; Cognition
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either daridorexant or placebo. Randomisation will be conducted using a variance minimisation procedure (Sella, Raz & Cohen Kadosh, 2021) to balance baseline sleep chronotype and gender across groups. Each participant will receive a single oral dose of daridorexant (50 mg) or placebo, followed by pupillometry and cognitive/emotional assessments approximately one hour post-dose. The study aims to examine the effects of dual orexin antagonism on aversive learning and cognition, is not designed as an efficacy or safety trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Data Collectors, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daridorexant (Experimental): Acute daridorexant (50mg)
  Interventions: Drug: Daridorexant 50 mg
- Placebo (Placebo Comparator): Inactive placebo comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Daridorexant 50 mg — Acute (single dose) daridorexant encapsulated in an opaque capsule. Oral administration. Daridorexant (brand name Quviviq) is FDA-approved for the treatment of insomnia in adults.
  Arms: Daridorexant
Other: Placebo — Lactose film-coated tablet will be encapsulated in an opaque capsule (identical to the experimental arm drug).
  Arms: Placebo

SUMMARY:
In this study, the investigators will examine the effects of blocking the orexin system on human behaviour and brain function using daridorexant, a medication that inhibits orexin activity. Orexin is a brain chemical involved in regulating sleep, emotion, motivation, and stress responses, which are often disrupted in mental health disorders. Healthy volunteers will be randomly assigned to receive a single dose of daridorexant or placebo in a double-blind design. Participants will then complete behavioural and cognitive tasks assessing emotional processing, aversive learning, and executive function. The study aims to clarify the role of orexin in emotional and cognitive processes relevant to conditions such as depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant, aged 18 to 30 years
* Willing and able to give informed consent for participation in the trial
* Able to follow study procedures as laid out in the participant information sheet
* Able to read and understand English
* Willing to avoid drinking alcohol, using recreational drugs, drinking grapefruit juice 24 hours before and after the study visit
* Willing to avoid driving or engaging in any activities requiring full alertness (e.g. cycling or operating heavy machinery) until the morning after the study visit day.
* Able to complete computer tasks without eye glasses even if uses correction regularly

Exclusion Criteria:

1. History of, receiving or seeking treatment for any sleep or circadian rhythm disorder or positive in screening questionnaires.
2. History of, receiving or seeking treatment for any clinically significant mental health condition (including but not limited to schizophrenia, psychosis, bipolar affective disorder, major depressive disorder, obsessive compulsive disorder, post-traumatic stress disorder) or positive in screening questionnaires.
3. History of, or current medical condition(s) which might increase the risk of oral administration of daridorexant, including:

   * ADHD requiring treatment with stimulants or other centrally-acting drugs
   * Neurological problems, including traumatic brain injury, epilepsy, Central Nervous System tumours or other severe neurological problems (e.g. Parkinson's disease; blackouts requiring hospitalisation)
   * Current Asthma, Chronic Obstructive Pulmonary Disease, emphysema or any medical condition that affects the lungs or breathing
   * Mild to severe hepatic impairment (Child-Pugh class A-C)
   * Severe renal disease
   * Severe gastrointestinal problems
   * History of, or current medical condition(s) which, in the opinion of the Investigator may interfere with the safety of the participant or the scientific integrity of the study
4. Pregnancy (as determined by urine pregnancy test taken during screening visit), intention to become pregnant or breastfeeding during the study or over the following six months.
5. Body mass index (BMI) below 18 or above 30kg/m2.
6. Current or past history of drug or alcohol dependency.
7. Use of recreational drugs or performance-enhancing drugs (e.g. cannabis, cocaine, amphetamines) within past three months.
8. Excessive caffeine consumption, i.e., consumption higher than 400mg a day of caffeine. This corresponds to more than 4 cups of brewed coffee, 6 espressos or filtered coffees, 9 cups of black tea, 10 cans of cola, or two "energy shot" drinks.
9. Smoking more than 5 cigarettes per day (or other nicotine replacement equivalent, including vaping on average more than 50 puffs a day).
10. Current or recent (past two months) use of any medication or medical devices (e.g. implanted neurostimulator) that affect brain function for the exception of contraceptives (pill, the Depo-Provera injection or the progesterone implant). This includes drugs that cause sedation (e.g. benzodiazepines, opioids, tricyclic antidepressants or sedative antipsychotics) or antihistamines.
11. Current use of any medications at risk of interaction with daridorexant; in particular:

    * strong or moderate CYP3A inhibitors (e.g. strong inhibitors - itraconazole, clarithromycin, ritonavir, grapefruit juice; moderate inhibitors - fluconazole, verapamil, diltiazem, erythromycin, ciprofloxacin, cyclosporine)
    * strong or moderate CYP3A inducers (e.g. of strong inducers - rifampicin, carbamazepine, St. John's wort; moderate inducers - bosentan, efavirenz, etravirine, modafinil)
    * Gastric pH-modifiers (e.g. famotidine and proton pump inhibitors such as omeprazole)
    * P-gp transporters (e.g. dabigatran, digoxin)
12. Inability to ingest up to 95mg of lactose.
13. Previous participation in any other drug study or sleep intervention study in the last three months.
14. Previous participation in any other study by the Psychopharmacology and Emotion Research lab (Department of Psychiatry, University of Oxford) or which uses the same computer tasks in the last 6 months
15. Participant is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pavlovian Aversive Learning Task Computational Parameter Estimates | 1-2 hours after single dose of drug or placebo.
  Change in the participant-specific parameter estimates produced by task model fitting.
Affective Go/No-Go Task Computational Parameter Estimates | 1-2 hours after single dose of drug or placebo.
  Change in the participant-specific parameter estimates produced by task model fitting.

SECONDARY OUTCOMES:
Pupilometry during Pavlovian Aversive Learning Task | 1-2 hours after single dose of drug or placebo.
  Changes in pupil size (dilation or constriction) in response to task stimuli
Pupilometry during Affective Go/No-Go Task | 1-2 hours after single dose of drug or placebo.
  Changes in pupil size (dilation or constriction) in response to task stimuli.
Salivary Alpha Amylase Levels | 1-2 hours after single dose of drug or placebo.
  Changes in Salivary Alpha Amylase Levels before, during and after Pavlovian Aversive Learning Task
Optimal choice selection during loss and reward conditions in Probabilistic Instrumental Learning Task (PILT) | 2-3 hours after single dose of drug or placebo.
  Optimal choice selection during loss and reward conditions in Probabilistic Instrumental Learning Task (PILT) in drug group compared with the placebo group
Accuracy of target selection on the Colour Change Detection Task | 2-3 hours after single dose of drug or placebo.
  Accuracy of target selection on the Colour Change Detection Task in pilosant group compared with the placebo group.
Accuracy of emotional labeling of facial expressions during the facial emotion recognition task | 2-3 hours after single dose of drug or placebo.
  Accuracy of emotion labels (e.g. disgusted face) assigned by participants to expressive faces during the facial emotion recognition task in drug group compared with the placebo group
Accuracy during categorisation of emotional words | 2-3 hours after single dose of drug or placebo.
  Accuracy to categorise positive and negative descriptor words
Accuracy during recall of emotional words | 2-3 hours after single dose of drug or placebo.
  Number of words accurately recalled
Pavlovian Aversive Learning Task Behavioural Performance | 1-2 hours after single dose of drug or placebo.
  Change in behavioural performance (response time; accuracy)
Affective Go/No-Go Task Behavioural Performance | 1-2 hours after single dose of drug or placebo.
  Change in behavioural performance (response time; accuracy)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Harmer, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data which has been fully de-identified may be shared with other academic and commercial organisations in the future, including those outside of the UK and the EU. Participants will be informed of this and specific consent to this is obtained within the Informed Consent Form.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: A few months after all data has been completed (ETA Oct 2026), unblinding has occurred (ETA Dec 2026), and all data analyses has been completed (Dec 2027).
Access Criteria: The data will be made publicly available. Access requests will not be required.
URL: https://osf.io/k6gmd/

REFERENCES:
- Available data/document: Study Protocol — https://osf.io/8mvn6
- Available data/document: Informed Consent Form — https://osf.io/5kuyn